CLINICAL TRIAL: NCT03983746
Title: Randomized Controlled Trial
Brief Title: Effect of Core Stability Exercises and Treadmill Training on Balance in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Saeed Alsakhawi, Lecturer, Faculty of Physical Therapy, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/ 013/001928
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Physical Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- traditional physical therapy program (control group) (Experimental): fifteen children with DS received a traditional exercises program with instructions to the children for 60 minutes aiming to improve posture control and balance
  Interventions: Device: core stability exercises and treadmill training exercises

INTERVENTIONS:
Device: core stability exercises and treadmill training exercises — Forty-five children with Down syndrome included in the study. The children aged 4-6 years, and they were equally divided randomly into three groups (A), (B) and (C). Group A received traditional physical therapy intervention strategies to facilitate the balance of participated children. Group (B) received same as the group (A), with additional core stability exercises training. Group (C) received same intervention strategies as group (A) in conjunction with a treadmill exercise program. The children's balance was evaluated using the Berg Balance Scale and the Biodex Balance System. Treatment sessions were for 60 min, thrice a week, for eight consecutive weeks.
  Other Names: traditional physical therapy program

SUMMARY:
Introduction: Core stability exercises and treadmill training play a crucial role in physical therapy interventions and have an effect on balance in children with Down syndromes (DS), whether core stability exercises or treadmill training has more effect on improve balance has not been investigated yet. The aim of the study was to investigate the effect of core stability training versus treadmill exercises on balance in children with Down syndrome. Methods: Forty-five children with Down syndrome included in the study. The children aged 4-6 years, and they were equally divided randomly into three groups (A), (B) and (C). Group A received traditional physical therapy intervention strategies to facilitate the balance of participated children. Group (B) received same as the group (A), with additional core stability exercises training. Group (C) received same intervention strategies as group (A) in conjunction with a treadmill exercise program. The children's balance was evaluated using the Berg Balance Scale and the Biodex Balance System. Treatment sessions were for 60 min, thrice a week, for eight consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to recognize commands given to them,
* Able to understand our verbal command and encouragement, and
* Able to stand and walk independently without repeated falling

Exclusion Criteria:

* Any neurological or musculoskeletal disorders (signs of epilepsy and instability of atlantoaxial joint),
* Any mobility disorders
* Any cardiac anomalies
* Any vision or hearing loss

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Functional Balance | 30 minutes
  The Biodex Balance System (BBS) is used to adjust the stability of a suspended circular force plate. The force platform has a maximum of twenty degrees tilt in any direction when completely un-stabilized and determines the stability of participant based on the variance of the platform from the center. The Berg Balance Scale is a clinical assessment of functional balance. It consists of fourteen functional tasks of increasing difficulty, and each scored on a scale ranging from 0 to 4 (task is performed independently=4; unable to complete the task=0). The maximum possible score is fifty-six which indicating no identifiable balance difficulties.
Overall Stability Index | 30 minutes
  The Biodex Balance System (BBS) is used to adjust the stability of a suspended circular force plate. The force platform has a maximum of twenty degrees tilt in any direction when completely un-stabilized and determines the stability of participant based on the variance of the platform from the center . The Berg Balance Scale is a clinical assessment of functional balance. It consists of fourteen functional tasks of increasing difficulty, and each scored on a scale ranging from 0 to 4 (task is performed independently=4; unable to complete the task=0). The maximum possible score is fifty-six which indicating no identifiable balance difficulties

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Cairo Governorate, Egypt